CLINICAL TRIAL: NCT06799442
Title: Dexmedetomidine Versus Fentanyl As Adjuvants to Erector Spinae Plane Block for Postoperative Analgesia Following Simple Nephrectomy: a Randomized Clinical Trial
Acronym: DEX/Fentanyl
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Bahgat Haleem Zaki, Resident physican, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX/Fentanyl ESPB Nephrectomy
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-09

CONDITIONS: Nephrectomy
Keywords: Postoperative pain relief
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients will be placed in lateral position with the surgical site upward. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. An echogenic needle needle will be inserted using an in-plane approach and craniocaudally direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.
  Group D patients: A total of 30 ml Bupivacaine 0. 25%+ 50 mic dexmedetomidine which is diluted to 2ml.
  Group F patients : A total of 30 ml Bupivacaine 0.25% + 100 mic fentanyl which is also diluted to 2 ml.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent anesthesiologist randomly divided the patients into 2 groups of 23 patients each using computer-generated random numbers dexmedetomidine group and fentanyl group (Group D and Group F). We discreetly placed the randomization results in envelopes until the end of the study. Both dexmedetomidine and fentanyl are colourless liquids, and they were digitally encoded after being diluted to 2 ml so that the researchers who are responsible for postoperative follow-up and data processing are blinded to the group allocation during the whole study period. All patients are also blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group dexmedetomidine (Active Comparator): Patients will be placed in lateral position with the surgical site upward. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. An echogenic needle needle will be inserted using an in-plane approach and craniocaudally direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.
  Group D patients: A total of 30 ml Bupivacaine 0. 25%+ 50 mic dexmedetomidine which is diluted to 2ml.
  Interventions: Procedure: Erector Spinae Plane Block; Drug: Dexmedetomidine
- Group fentanyl (Active Comparator): Patients will be placed in lateral position with the surgical site upward. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. An echogenic needle needle will be inserted using an in-plane approach and craniocaudally direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.
  Group F patients : A total of 30 ml Bupivacaine 0.25% + 100 mic fentanyl which is also diluted to 2 ml.
  Interventions: Procedure: Erector Spinae Plane Block; Drug: fentanyl

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Patients will be placed in lateral position with the surgical site upward. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. An echogenic needle needle will be inserted using an in-plane approach and craniocaudally direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.
Drug: Dexmedetomidine — 50 mic dexmedetomidine which is diluted to 2ml.
  Arms: Group dexmedetomidine
Drug: fentanyl — 100 mic fentanylwhich is also diluted to 2 ml.
  Arms: Group fentanyl

SUMMARY:
The aim of this clinical trial is to compare the time to first analgesic request between dexmedetomidine and fentanyl as adjuvants in erector spinae plane block in patients undergoing simple nephrectomy .

• Secondary outcome Pain scores; Numerical Rating Scale (NRS) at rest and when coughing [at 1, 2, 4, 8, 16 and 24 hours postoperatively.] The total opiod dose in the first 24 hours postoperatively. Duration of analgesia is defined as duration between block administration and time of first analgesic request.

Any adverse effects related to anesthesia or the technique. Incidence of Postoperative nausea & vomiting . Block related complication during and after block procedure till 24hours postoperatively (local anesthetic systemic toxicity, pneumothorax and vascular puncture during block procedure).

Intraoperative haemodynamics parameters MAP ,HR , co2 and SP O2 . Postoperative haemodynamics parameters MAP , HR and SP O2 [at 1, 2, 4, 8, 16 and 24 hours postoperatively. ]

DETAILED DESCRIPTION:
An independent anesthesiologist randomly divided the patients into 2 groups of 23 patients each using computer-generated random numbers dexmedetomidine group and fentanyl group (Group D and Group F). We discreetly placed the randomization results in envelopes until the end of the study. Both dexmedetomidine and fentanyl are colourless liquids, and they were digitally encoded after being diluted to 2 ml so that the researchers who are responsible for postoperative follow-up and data processing are blinded to the group allocation during the whole study period. All patients are also blinded to the group allocation.

A)Anaesthesia induction:

Standard monitoring procedures will include pulse oximetry, electrocardiography, and noninvasive arterial pressure prior to anesthetic induction. All patients will be premedicated with intravenous (i.v.) midazolam 1-2 mg and antibiotic prophylaxis, according to the hospital's protocol. Anesthesia will be induced with intravenously (IV)-administered propofol 2 mg/kg, fentanyle 1 mic kg following which endotracheal intubation will be facilitated by atracurium 0.5 mg / kg. Anesthesia will be maintained with oxygen, air, and isoflurane using controlled ventilation with closed circuit in order to ensure normocarbia. Regular doses of atracurium 0.25 mg / kg will be given every 20 minutes to ensure proper muscle relaxation. After positioning the patient of the surgery, patients will receive their intervention according to group allocation under sterile conditions.

B)Intervention:

Erector Spinae Plane Block:

Patients will be placed in lateral position with the surgical site upward. A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. An echogenic needle needle will be inserted using an in-plane approach and craniocaudally direction. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.

Group D patients: A total of 30 ml Bupivacaine 0. 25%+ 50 mic dexmedetomidine which is diluted to 2ml.

Group F patients : A total of 30 ml Bupivacaine 0.25% + 100 mic fentanyl which is also diluted to 2 ml.

Intraoperativeely

The following parameters will be monitored intraoperatively :

HR and MAP and SpO2 and CO2 will be documented at induction, intubation, surgical incision and every 15 min. till the end of surgery.

* Perflgan 1gm and Ondansetron 0.1 mg/kg will be given at the end of the procedure to all patients.
* Neuromuscular blockade will be reversed with neostigmine and atropine at the end of the procedure.

Post operative

* Postoperative pain will be assessed using an 11-point (0=no pain and 10=worst pain) numeric rating scale (NRS). NRS for pain at rest and when coughing will be assessed serially at 1, 2, 4, 8, 16 and 24 h after surgery. The assessor and the patients will be unaware of the type of intervention received.
* Rescue analgesics will be administered when NRS ≥4 or when the patient complains of pain. In the firm of the nalbuphine 0.1 mg /kg
* Time for first analgesic request will be recorded. The duration of analgesia will be evaluated as the time from block administration to the time of first analgesic. Total doses of rescue analgesics required in the first 24 h will be recorded.
* The presence of postoperative nausea and vomiting during the first 24 h will be recorded. Postoperative nausea or vomiting will be treated with 0.1 mg/kg of ondansetron. If the patient did not respond to ondansetron, then dexamethasone 8 mg or metoclopramide 10 mg will be given IV. Occurrence of any complications such as haematoma, bleeding, local anesthetic systemic toxicity, pneumothorax and allergic reactions will also be observed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old Both sex patients who are American society of Anesthesiologists class I or

Exclusion Criteria:

* Patient's refusal.
* body mass index (BMI) ≥40 kg/m2.
* Local infection at site of block.
* Spine deformities
* History of hypersensitivity to the drugs being evaluated
* Inability to comprehend postoperatively the pain assessment scale/neuropsychiatric disorders.
* Chronic use of opioids and opioid addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the time to first analgesic request | 24 hours
  To compare the time to first analgesic request between dexmedetomidine and fentanyl as adjuvants in erector spinae plane block in patients undergoing simple nephrectomy .

SECONDARY OUTCOMES:
Pain scores | 24 hours
  Numerical Rating Scale (NRS) when coughing
The total opiod dose | 24 hours
  The total opiod dose postoperatively
Duration of analgesia | 24 hours
  Duration of analgesia is defined as duration between block administration and time of first analgesic request.
Postoperative nausea & vomiting | 24 hours
  Incidence of Postoperative nausea & vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Moamen Mostafa Makkey, Doctor, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Waloejo CS, Musalim DAP, Budi DS, Pratama NR, Sulistiawan SS, Wungu CDK. Dexmedetomidine as an Adjuvant to Nerve Block for Cancer Surgery: A Systematic Review and Meta-Analysis. J Clin Med. 2024 May 28;13(11):3166. doi: 10.3390/jcm13113166. PMID 38892876
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Adhikary SD, Bernard S, Lopez H, Chin KJ. Erector Spinae Plane Block Versus Retrolaminar Block: A Magnetic Resonance Imaging and Anatomical Study. Reg Anesth Pain Med. 2018 Oct;43(7):756-762. doi: 10.1097/AAP.0000000000000798. PMID 29794943
- [Background] De la Cuadra-Fontaine JC, Concha M, Vuletin F, Arancibia H. Continuous Erector Spinae Plane block for thoracic surgery in a pediatric patient. Paediatr Anaesth. 2018 Jan;28(1):74-75. doi: 10.1111/pan.13277. No abstract available. PMID 29226529
- [Background] Finneran JJ 4th, Gabriel RA, Khatibi B. Erector Spinae Plane Blocks Provide Analgesia for Breast and Axillary Surgery: A Series of 3 Cases. Reg Anesth Pain Med. 2018 Jan;43(1):101-102. doi: 10.1097/AAP.0000000000000695. No abstract available. PMID 29261601
- [Background] Bonvicini D, Giacomazzi A, Pizzirani E. Use of the ultrasound-guided erector spinae plane block in breast surgery. Minerva Anestesiol. 2017 Oct;83(10):1111-1112. doi: 10.23736/S0375-9393.17.12015-8. Epub 2017 May 11. No abstract available. PMID 28492298
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Capdevila X, Moulard S, Plasse C, Peshaud JL, Molinari N, Dadure C, Bringuier S. Effectiveness of Epidural Analgesia, Continuous Surgical Site Analgesia, and Patient-Controlled Analgesic Morphine for Postoperative Pain Management and Hyperalgesia, Rehabilitation, and Health-Related Quality of Life After Open Nephrectomy: A Prospective, Randomized, Controlled Study. Anesth Analg. 2017 Jan;124(1):336-345. doi: 10.1213/ANE.0000000000001688. PMID 27918333
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Misiolek H, Cettler M, Woron J, Wordliczek J, Dobrogowski J, Mayzner-Zawadzka E. The 2014 guidelines for post-operative pain management. Anaesthesiol Intensive Ther. 2014 Sep-Oct;46(4):221-44. doi: 10.5603/AIT.2014.0041. No abstract available. PMID 25293474
- [Background] Sharma V, Margreiter M. Partial nephrectomy: is there still a need for open surgery? Curr Urol Rep. 2013 Feb;14(1):1-4. doi: 10.1007/s11934-012-0297-2. PMID 23233109
- [Background] Sahin A, Baran O. Effect of ultrasound-guided erector spinae plane block on post-surgical pain in patients undergoing nephrectomy: a single-center, randomized, double-blind, controlled trial. J Int Med Res. 2022 Mar;50(3):3000605221086737. doi: 10.1177/03000605221086737. PMID 35301896